CLINICAL TRIAL: NCT06094374
Title: Unveiling the Digital Phenotype: A Protocol for a Prospective Study on Physical Activity Behavior in Community-dwelling Older Adults
Brief Title: Unveiling the Digital Phenotype of PA Behavior
Acronym: MIADP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: PXL University College (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Other Study IDs: MIADP
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Physical Activity - Digital Phenotyping - Activity Tracking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community Dwellling Healthy Older Adults: * 65 years or older
  * able to give informed consent
  * community dwelling
  * no severe illness (neurological, cardiovascular, respiratory, metabolic, cognitive disorder)
  * dutch language profiency
  Interventions: Behavioral: observation of physical activity behavior

INTERVENTIONS:
Behavioral: observation of physical activity behavior — An observational study will be conducted to gather data on multiple levels aiming to identify diverse digital phenotypes related to PA behavior among community-dwelling older adults.
  A hybrid approach will be employed, combining both cross-sectional and longitudinal data collection methods. The overall aim is to employ data analysis to identify patterns of PA - behavior (referred to as phenotypes) and to pinpoint prognostic factors that affect PA outcomes.
  This integrated strategy will be complemented by four distinct measurement approaches, ensuring a comprehensive assessment of the research objectives. These measurement approaches include:self-reporting, clinical, ecological momentary and time series assessment.

SUMMARY:
Observational data from healthy adults aged 65+ will be collected through cross-sectional and longitudinal methods to analyze physical activity patterns, identifying digital phenotypes. Measurements include self-reports, clinical assessments, and EMA, with statistical analysis using multivariate regression and time series analysis, and a neural network if needed to find digital phenotypes related to physical activity in older adults.

DETAILED DESCRIPTION:
Observational data will be collected in healthy older adults aged 65 or above combining both cross-sectional and longitudinal data collection methods to analyze patterns of PA behavior and identify prognostic factors affecting PA outcomes in order to identify digital phenotypes related to PA.

The measurements are based on the Behavioral Change Wheel and include self-reporting assessments, clinical assessments for cross-sectional data collection and ecological momentary assessment (EMA) as well as time series data collection for longitudinal data. The statistical analysis will involve multivariate regression analysis and time series analysis, with a Bonferroni correction to account for multiple comparisons. A machine learning algorithm is used due to the complexity of the data. If no suitable model is found, a neural network will be used to determine digital phenotypes related to PA behavior in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 65 years of older
* Participants are competent to give informed consent
* Participants are able to actively participate in the study
* Participants are community-dwelling (living independent at home or in a service apartment)
* Without a severe illness
* Dutch language proficiency as native speaker

Exclusion Criteria:

* Current neurological disorder such as Parkinson's disease, multiple sclerosis, cerebrovascular accident, …
* Current cardiovascular disorder such as stroke, acute myocardial infarct, coronary artery bypass grafting, percutaneous coronary intervention less than 5 years ago
* Current respiratory disorder, such as chronic obstructive pulmonary disease, pneumonia, pulmonary fibrosis, asthma, …
* Current severe metabolic disorder, such as diabetes type 1 and 2, severe osteoporosis, …
* Current severe cognitive disorders, such as Alzheimer's disease, vascular dementia, Lewy Body dementia, frontotemporal dementia,

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Healthy Community Dwelling older adults aged 65 years or more
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Digital phenotypes of PA | 14 days
  Patterns of physical activity behavior

CONTACTS AND LOCATIONS:
Overall Officials: Kim Daniels, MS, Principal Investigator — PXL University College of Applied Sciences and Arts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Daniels K, Vonck S, Robijns J, Spooren A, Hansen D, Bonnechere B. Characterising physical activity patterns in community-dwelling older adults using digital phenotyping: a 2-week observational study protocol. BMJ Open. 2025 May 24;15(5):e095769. doi: 10.1136/bmjopen-2024-095769. PMID 40413040